CLINICAL TRIAL: NCT04622605
Title: Hydrus Microstent and Lens Extraction for the Treatment of Primary Angle-Closure Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Eye Institute (Industry)
Collaborators: Ivantis, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Edward T. Ang, Principal Investigator, Asian Eye Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Primary Angle Closure Glaucoma; Primary Angle Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Cataract extraction and intraocular lens placement with combined placement of glaucoma microstent
  Interventions: Device: Trabecular bypass and Schlemm's canal stent

INTERVENTIONS:
Device: Trabecular bypass and Schlemm's canal stent — ab interno Microstent placement after cataract surgery
  Other Names: Hydrus Microstent

SUMMARY:
This study is a prospective evaluation of the Hydrus Microstent for the treatment of Primary Angle Closure (PAC) and Primary Angle Closure Glaucoma (PACG) with adjunctive cataract. A total of 20 subjects will be successfully treated with one Hydrus device after completion of cataract extraction with phacoemulsification followed by IOL replacement (HMS cohort), and 10 eyes will be treated with phacoemulsification cataract extraction and IOL replacement only (PCS group). Since cataract surgery is standard of care for this condition, eligible fellow eyes from the HMS cohort may be enrolled into the PCS group. To avoid selection bias in this non-randomized study, the first 20 consecutive qualifying subjects will be treated with Hydrus and the next 10 consecutive qualifying eyes will be treated with cataract surgery only.

DETAILED DESCRIPTION:
The objective of this study is to assess the effectiveness of the Hydrus Microstent for lowering intraocular pressure in patients with PAC or PACG. The addition of the Hydrus is expected to lower IOP and medication dependency, and thus reduce the risk of progression of glaucoma. The PCS group will provide a control group to assess the magnitude of the Hydrus treatment effect on IOP, medications, and safety.

Upon successfully meeting the study inclusion/exclusion criteria at both the screening and baseline visits, the subject will be scheduled for surgery. Follow up will be continued for 1 year post surgery, and will include assessments of the subject's IOP, ocular health, and visual acuity status. Visits will be conducted at 1, 7, 30, 90, 180, and 365 days.

A 20% drop in IOP in response to therapy is considered clinically meaningful. The study treatment will be considered successful if a patient can obtain this response in IOP using the same or a fewer number of medications as pre-operative baseline.

ELIGIBILITY:
Inclusion Criteria:

Pre-Operative Inclusion Criteria

1. Male and Female patients at least 40 years of age.
2. An operable age-related cataract with visual impairment or glare, eligible for phacoemulsification.
3. Subjects with diagnosed primary angle-closure (PAC; defined as appositional or synechial irido-trabecular contact of 90 degrees or more on gonionscopy) OR primary angle-closure glaucoma (PACG; defined as PAC with documented glaucomatous optic neuropathy and/or reproducible glaucomatous visual field defect), and on > or = 1 glaucoma medication with IOP > or = 21mmHg at both preoperative visits.
4. PAC or PACG subjects that are newly diagnosed, or unmedicated (newly diagnosed or non-compliant patient not using medication for > 30 days), with IOP > or = 24mmHg at both preoperative visits.

The subject is able to understand the requirements of the study and is willing to provide written informed consent, follow study instructions, and comply with all study procedures.

Intraoperative Inclusion Critera

1. An intact and centered capsulorhexis.
2. An intact posterior capsular bag.
3. A well-centered IOL implant placed in the capsular bag.
4. A clear view and visualization of the angle with direct gonioscopy.
5. No evidence of zonular dehiscence/rupture (uncomplicated cataract extraction)

Exclusion Criteria:

1. Pseudophakia in the intended study eye
2. All forms of glaucoma other than primary angle-closure (i.e. all open-angle glaucoma including primary open-angle, pseudoexfoliative, or pigmentary glaucoma; neovascular, uveitic, traumatic, steroid induced, lens induced, or glaucoma associated with increased episcleral venous pressure; congenital or developmental glaucoma).
3. Secondary angle-closure glaucoma
4. Advanced glaucoma, defined as visual field mean deviation worse than -15 dB, or cup-to-disc ration > or = 0.9.
5. Visual field depression within the central 5 degrees of fixation, on pattern deviation probability plot.
6. Eyes with an anticipated need for incisional glaucoma surgery (e.g. trabeculectomy or tube shunt) within the 12-month follow-up period.
7. Central corneal thickness >620 or <490 microns.
8. Axial length < or = 19 mm (nanophthalmos).
9. Previous incisional glaucoma surgery in the study eye, including trabeculectomy, tube shunt, and non-penetrating procedures such as deep sclerectomy, viscocanalostomy or canaloplasty.
10. Plateau iris syndrome.
11. History of complicated intraocular surgery.
12. Previous MIGS surgery in the study eye.
13. Proliferative diabetic retinopathy.
14. Previous surgery for retinal detachment.
15. Clinically significant corneal dystrophy (e.g. Fuch's Dystrophy).
16. Best-corrected visual acuity in the fellow eye worse than 20/200.
17. Previous corneal surgery.
18. Previous refractive surgery.
19. Degenerative visual disorders such as exudative age-related macular degeneration.
20. Clinically significant ocular inflammation or infection within thirty days prior to screening.
21. Uncontrolled systemic disease that in the opinion of the investigator would put the subject's health at risk and/or prevent the subject from completing all study visits.
22. Pregnant or nursing females.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Reduction in IOP | 12 months
  Proportion of subjects with > or = 20% reduction of IOP while maintaining the same or fewer number of glaucoma medications compared with baseline, measured by Goldmann applanation tonometry

SECONDARY OUTCOMES:
Change in IOP | 12 months
  Change in IOP compared to baseline IOP regardless of the number of glaucoma medications

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Eye Institute, Makati City, National Capital Region, Philippines